CLINICAL TRIAL: NCT03484598
Title: Clinical Utility of the SPEAC® System: A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS-1.5-01.2018
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SPEAC Treatment Arm (Experimental): All study participants will be provided with a SPEAC System to use in their home environment.
  Interventions: Device: SPEAC System

INTERVENTIONS:
Device: SPEAC System — A lightweight, non-invasive monitor that is placed on the belly of the biceps muscles to analyze surface electromyography (sEMG) signals that may be associated with generalized tonic-clonic (GTC) seizures. It provides an alarm to alert caregivers of unilateral, appendicular, tonic extension that could be associated with a GTC seizure. The System records and stores sEMG data for subsequent review by a trained healthcare professional.
  Other Names: Brain Sentinel Seizure Monitoring and Alerting System

SUMMARY:
The primary objective is to collect preliminary data related to the clinical utility of the SPEAC System in patients with a history of motor seizures. This trial is primarily an observational investigation. This protocol describes a series of observational case studies. Each case study is intended to be interpreted independent from the other case studies. Self-reported seizure frequency will be compared to observed seizure frequency using the SPEAC System.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a reported history of motor seizures (epileptic or not or unknown) with upper extremity motor involvement.
* The subject's first reported seizure must be within the last 5 years.
* Male or Female between the ages 22 and 99.
* If female and of childbearing potential, subject must agree to not become pregnant during the trial.
* Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments.
* Subject or Primary Caregiver must be competent to follow all study procedures.
* Subject must be willing to use the Seizure Monitoring and Alerting System for a long period of time (up to 90 days), for a minimum of 30 hours/ week.

Exclusion Criteria:

* The subject cannot be pregnant, or nursing.
* The subject cannot be sensitive or allergic to adhesives or tapes.

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Compare Seizure Frequency | 1 year
  We will compare self-reported seizure frequency to the seizure frequency measured by the SPEAC System.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The University of South Florida, Tampa, Florida
  - Austin Epilepsy Care Center, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No